CLINICAL TRIAL: NCT07362160
Title: Evaluating the Clinical Performance of a Novel Clear Orthodontic Expander Versus Hyrax: A Randomized Clinical Trial
Brief Title: Clear Orthodontic Expander Versus Hyrax
Acronym: COE-Hyarx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Noor Falah Kadhim Al-Khawaja, postgraduate/PhD student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1158425; 1158 (Other: College of Dentistry / University of Baghdad)
Record Dates: First submitted 2026-01-12; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Malocclusion; Narrow Maxilla
Keywords: clear expander; hyrax; clinical trial; adolescent; thermoplastic material
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: hyrax expander clear orthodontic expander
Who Masked: Participant, Outcomes Assessor
Masking Description: As the study will be conducted in different clinics, all data collection and measurement will be completed with the investigator being masked to the allocation groups, though blinding of the operator will not be possible due to the appliance design/shape difference, and for the cleaning methods, blinding will be applied for the bacteriological specialist, and for the outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New clear expander (Experimental): After obtaining the 3D-printed maxillary dental cast, a 2 mm PETG (rigid) thermoforming material (Leone® S.p.A., Florence, Italy) will be adapted separately to the maxillary cast using a pressure molding vacuum machine. The clear appliance will then be trimmed and finished. Depending on the degree of maxillary constriction, a Leone® Standard or universal expansion screw (Leone® S.p.A.,Florence, Italy) measuring 6-9 mm will be incorporated into the appliance and positioned in the midline of the maxillary cast after splitting the appliance midpalatally embedded in acrylic composed from Methyl methacrylate monomer and Methyl methacrylate polymer Orthocryl® liquid (monomer), and Orthocryl® EQ-powder (polymer) (Dentaurum GmbH & Co. KG, Ispringen, Germany)
  Interventions: Device: New clear expander
- Hyrax expander (Experimental): After obtaining the 3D-printed maxillary dental cast, patients will be treated with a Hyrax expander using a rapid expander from Leone® S.p.A., Florence, Italy, cemented in the upper first premolars and first molars. If the first premolars had not yet erupted, the Hyrax expander will be cemented in the upper first permanent molars only.
  Interventions: Device: Hyrax expander

INTERVENTIONS:
Device: New clear expander — All patients with a clear expander will be instructed to wear the appliance 24 hours a day, except during eating and cleaning. The expander will be activated twice daily (0.2 mm per turn). Patients will be provided with an instruction brochure and advised to use a reminder to ensure compliance. The expansion will continue until the desired amount of the maxillary arch expansion occurs when the maxillary first molars' palatal cusps occlude the lingual side of the mandibular first molar buccal cusps to overcome the expected relapse due to the elasticity of the palatal soft tissue.
  Arms: New clear expander
Device: Hyrax expander — The activation protocol for the Hyrax expander will be the same in all patients, twice daily (0.2 mm per turn). The expansion will continue until the desired amount of the maxillary arch expansion occurs when the maxillary first molars' palatal cusps occlude the lingual side of the mandibular first molar buccal cusps to overcome the expected relapse due to the elasticity of the palatal soft tissue.
  Arms: Hyrax expander

SUMMARY:
This study will be conducted to evaluate the effectiveness of a clear expander fabricated from 2-mm biocompatible polyethylene terephthalate glycol (PETG) thermoforming material integrated with an expansion screw in achieving dental and skeletal expansion in adolescent patients, compared with the conventional Hyrax expander.

DETAILED DESCRIPTION:
This will be a multicenter randomize clinical trial with two-arm parallel groups, and will be conducted at the Department of Orthodontics, College of Dentistry, University of Baghdad, as well as different specialized dental centers affiliated with the Iraqi Ministry of Health, and some private clinics.

The sample size will be calculated based on previous studies with similar aim to measure the skeletal expansion. A minimum sample size of 17 patients was required, and in order to account for a 15% dropout, a total of 20 patients will be recruited for each group (new clear expander and hyrax expander). The amount of 2.5 mm or greater of maxillary sutural opening will be considered clinically effective.

Two randomizations will be employed, one for the expander type and the other for the cleaning method of the new expander, a computer random generator will be used to develop a simple randomization with an equal allocation ratio (1:1) and without stratification.

Data Collection and Measurements will be include, CBCT evaluation, Intraoral scan of the maxillary arch evaluation, overjet and overbite, CBCT-derived cephalometric images will be used to measure the maxillary mandibular plane angle, Microbial evaluation after using two different methods for cleaning the new clear expander and at the end of the treatment, the patient will be asked to fill out a questionnaire about the treatment, giving information about their experience and satisfaction during treatment.

Data will be analyzed using the Statistical Package for Social Sciences for Windows, version 26.0, including Descriptive Statistics 9numbers, frequencies, percentages, mean, median, and standard deviations), Reliability Statistics (an intraclass correlation coefficient), and Inferential Statistics (Levene's test, Shapiro Wilk test, Paired samples t-test and Independent samples t-test).

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age at the start of treatment will range from 10-14 years.
2. Unstable unilateral or bilateral posterior crossbite due to maxillary constriction.
3. The first molars are fully erupted.
4. Good oral health free from caries and periodontal problems at the start of treatment.
5. Good general health.

Exclusion Criteria:

1. Patients with a vertical growth pattern.
2. Patients with obvious facial asymmetry.
3. Patients with orofacial cleft.
4. Patients with previous orthodontic treatment.
5. Patients with bad oral habits.
6. Patients with active periodontal disease.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
CBCT evaluation | pre-treatment (T0) and immediately post-treatment (T1) around one to two months
  Skeletal and dentoalveolar measurements will be assessed using cone-beam computed tomography (CBCT). Skeletal measurements will include nasal width, midpalatal suture gap, and palatal height, measured in millimeters (mm). Dentoalveolar measurements will include vertical dental heights and maxillary width measured in millimeters (mm), as well as dental inclination measured in degrees (°). All measurements will be obtained from CBCT images using dedicated three-dimensional imaging analysis software.

SECONDARY OUTCOMES:
Intraoral scan of the maxillary arch evaluation | pre-treatment (T0) and post-treatment (T1) around one to two months
  Maxillary transverse dental measurements will be assessed using a digital intraoral scan. The parameters evaluated will include intercanine width, interpremolar width, intermolar width, and intermolar transpalatal width, all measured in millimeters (mm) using three-dimensional digital dental model analysis software.
Clinical evaluation | pre-treatment (T0) and immediately post-treatment (T1) around one to two months
  Overjet and overbite will be evaluated clinically using a calibrated orthodontic ruler, with measurements recorded in millimeters (mm).
Cephalometric analysis | pre-treatment (T0) and immediately post-treatment (T1) around one to two months
  CBCT-derived cephalometric images will be used to measure the maxillary mandibular plane angle in degrees (°) to evaluate the vertical relationship using cephalometric analysis software.
Microbial evaluation | after one month.
  Patients will be allocated into two groups according to the cleaning method: brushing with a toothbrush and aligner foam (China) or using Efferdent cleaning tablets (USA). Biofilm samples will be collected using sterile swabs with Amies transport medium (Boen Healthcare Co., Ltd., China). The outcome measure will be bacterial biofilm accumulation, assessed by bacteriological analysis based on bacterial colony counting, expressed as colony-forming units per milliliter (CFU/ml).
Patient satisfaction with the appliance | around one to two months
  At the end of treatment, patient-reported experience and satisfaction will be assessed using a structured questionnaire. Responses will be recorded as questionnaire scores using a 3-point Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yassir A Yassir, Ph.D. (UK), Study Chair — University of Baghdad
Locations (1):
- University of Baghdad/Collage of Dentistry, Baghdad, Al-Rusafa, Bab Al-moadham, Iraq

IPD SHARING:
Plan to Share IPD: No